CLINICAL TRIAL: NCT03269240
Title: A Comparative Study of Simulation-based Low-dose High Frequency (LDHF) Plus Mobile Mentoring (m-Mentoring) Versus Traditional Group-based Training Approaches Among Maternal and Newborn Healthcare Providers in Ebonyi and Kogi States, Nigeria
Brief Title: Simulation-based Low-dose High Frequency (LDHF) Plus Mobile Mentoring (m-Mentoring) Study in Nigeria
Acronym: LDHF-Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00007196
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Training; Capacity Building; Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Clinical Competence

STUDY DESIGN:
Intervention Model Description: Cluster randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The assessors will blinded with respect to which study arm the participants (health care workers) were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDHF plus m-Mentoring (Experimental): Participants will undergo pre-training assessment comprising multiple-choice questions and objective structured clinical examination (OSCE) using manikins. Training is divided into two 4-day "low-dose" sessions at the health facility or onsite training. Pre-training and immediate post-training assessments results will be compared. A score of ≥80% is acceptable competence (pass). During the one-month intervals between training sessions, participants practice using manikins to reinforce their competencies through simulation-based practices, facilitated by facility-based trained Peer Practice Coordinators (PPCs). The PPCs will also receive structured, monthly half-hour mentoring calls that will provide remote support, answering questions, providing guidance and reinforcing key messages. Acquisition of knowledge and clinical skills is measured.
  Interventions: Behavioral: Acquisition of Knowledge and clinical skills; Other: Onsite training
- Traditional training (Active Comparator): The health providers will receive the same content of training in eight days, Off-site training, the way it's currently done in Nigeria. Both theoretical and practical through use of manikins - simulation. No reinforcement and further practice will take place once the participants are back in their work stations. Acquisition of knowledge and clinical skills is measured.
  Interventions: Behavioral: Acquisition of Knowledge and clinical skills; Other: Off-site training

INTERVENTIONS:
Behavioral: Acquisition of Knowledge and clinical skills — LDHF is a novel training approach that is being compared to the traditional training approach
Other: Onsite training — Participants are training at their health facilities
  Arms: LDHF plus m-Mentoring
Other: Off-site training — Participants from different health facilities are gathered together in a central location for training, away from their workplaces
  Arms: Traditional training

SUMMARY:
The aim of this study is to compare the effectiveness and cost of a simulation-based low dose high frequency (LDHF) plus m-Mentoring training versus the traditional group-based training approaches in improving knowledge and skill in maternal and newborn care and to determine trainees' satisfaction with the approaches in Ebonyi and Kogi states.

The specific objectives are to:

1. Compare knowledge and skill learning outcomes between the two groups of birth attendants trained through the simulation-based LDHF/m-Mentoring versus group-based training approaches in Kogi and Ebonyi states over 12-months.
2. Assess the trainees' satisfaction with a simulation-based LDHF/m-Mentoring and group-based training approaches in improving skills of birth attendants in the selected facilities in Kogi and Ebonyi state over 12-months.
3. Determine the cost and cost-effectiveness of LDHF/m-Mentoring and group-based training approaches in improving skills of birth attendants in the selected facilities in Kogi and Ebonyi state over 12-months.

DETAILED DESCRIPTION:
Simulation-based low dose high frequency (LDHF) training has emerged as a new strategy for delivering key content and improving the competencies of health workers. In facility-based driven simulation-based LDHF trainings, providers are not removed from clinical practice for the extended periods of time, and a heavy emphasis is placed on simulation with practice and feedback.

The Maternal and Child Survival Program (MCSP) in Nigeria is working in selected health facilities in Ebonyi and Kogi States to improve the quality of care received by mothers and newborns on the day of birth using high-impact evidence-based lifesaving interventions. The simulation-based LDHF/m-Mentoring evaluation comparing it to the traditional group-based training will contribute to the body of knowledge on this approach.

The study design is cluster randomized control trial. Sixty (60) health facilities will be selected from the list of 120 facilities which are supported by MCSP and randomized to intervention and control group. Selection will be based on caseload, level of service delivery, and ownership. Thereafter, these will be randomly assigned to simulation-based LDHF/m-Mentoring Group (intervention arm) or Group-Based Training Group (control arm).

ELIGIBILITY:
Inclusion Criteria:

1. Must give informed consent to participate in the study;
2. Must have spent at least six months in maternal and/or newborn care services;
3. Must be providing services related to maternal and newborn health in selected health facilities at the time of the interview;
4. Must be available to participate in the training from the beginning to the end; and
5. Must have had pre-service training not incorporating simulation-based LDHF approach from accredited medical schools, schools of nursing/midwifery or health technology.

Exclusion Criteria:

1. Decides to opt out / declines to participate.
2. Has had prior training using the simulation-based LDHF approach.
3. Provides services related to maternal and newborn health more than one health facility selected as part of intervention or comparison group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2016-09-17 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Percent change in competency in basic obstetric and emergency care between the groups | 3 months
  Proportion of competent providers who retain clinical competency skills 3 months post-training

SECONDARY OUTCOMES:
Comparison of retention of skills between the two study arms | 12 months
  Proportion of service providers who retain clinical competency skills after 12 months
Level of satisfaction of service providers | 12 months
  Proportion of service providers who are satisfied with the training approach
Comparison of cost-effectiveness of the two approaches | 12 months
  Cost-effectiveness of LDHF/m-Mentoring compared to group-based training approaches in improving skills of birth attendants in the selected facilities in Kogi and Ebonyi states.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Otolorin, Principal Investigator — Jhpiego

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol will be shared through publication in a peer-reviewed journal.
  De-identified participant data will be submitted to a data repository in accordance with the USAID policy where other researchers will have access.

REFERENCES:
- [Derived] Ugwa E, Kabue M, Otolorin E, Yenokyan G, Oniyire A, Orji B, Okoli U, Enne J, Alobo G, Olisaekee G, Oluwatobi A, Oduenyi C, Aledare A, Onwe B, Ishola G. Simulation-based low-dose, high-frequency plus mobile mentoring versus traditional group-based trainings among health workers on day of birth care in Nigeria; a cluster randomized controlled trial. BMC Health Serv Res. 2020 Jun 26;20(1):586. doi: 10.1186/s12913-020-05450-9. PMID 32590979
- [Derived] Ugwa E, Otolorin E, Kabue M, Ishola G, Evans C, Oniyire A, Olisaekee G, Onwe B, LeFevre AE, Bluestone J, Orji B, Yenokyan G, Okoli U. Simulation-based low-dose, high-frequency plus mobile mentoring versus traditional group-based training approaches on day of birth care among maternal and newborn healthcare providers in Ebonyi and Kogi States, Nigeria; a randomized controlled trial. BMC Health Serv Res. 2018 Aug 13;18(1):630. doi: 10.1186/s12913-018-3405-2. PMID 30103761